CLINICAL TRIAL: NCT03437681
Title: Tissue-specific Effects of Insufficient Sleep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-0533
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Sleep; Blood Sugar

STUDY DESIGN:
Intervention Model Description: The project is a within-subject consecutive design examining 18 healthy individuals after baseline and after 4 nights of insufficient sleep.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insufficient sleep (Experimental): Each participant will receive 4 nights of insufficient sleep.
  Interventions: Behavioral: Insufficient sleep

INTERVENTIONS:
Behavioral: Insufficient sleep — Four days of insufficient sleep

SUMMARY:
This study plans to learn more about how sleep loss impacts the way the body responds to sugar. This work will have important implications for development of treatments and countermeasures for people who are not able to get enough sleep for various reasons.

DETAILED DESCRIPTION:
Participants will stay in the hospital for 6 days and will not be able to leave. Sleep habits will be measured for 7 days before the study. A research diet that is designed to maintain weight will be provided for 3 days before the study and during the study. Multiple tests will be performed, including metabolic testing and muscle and fat biopsies, both when participants first arrive and have had normal sleep and again after 4 nights of only 5 hours time in bed. The visit takes place at the Clinical Translational Research Center (CTRC) at the University of Colorado Denver, Anschutz Medical campus. It will take approximately 2 weeks to complete this study.

ELIGIBILITY:
Inclusion criteria:

1. Healthy, lean participants.
2. No regular physical activity (<20 minutes/day). No exercise will be allowed for 3 days prior to study start.
3. Habitual sleep duration between 7-9.25h. Subjects must also be willing and able to keep a 9h time-in-bed schedule for 1 week prior to study admission.
4. Potential subjects must have lived at Denver altitude or higher for at least 3 months to inpatient study.

Exclusion Criteria:

1. Current or history of any clinically significant medical, psychiatric, or sleep disorder.
2. Use or history of any drugs, medications, supplements, caffeine, and alcohol.
3. Current or history of shiftwork in six months prior to laboratory study.
4. Travel more than one time zone in three weeks prior to laboratory study.
5. Blood donation in the 30 days prior to inpatient study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity | One week
  Insulin sensitivity measured by hyperinsulinemic euglycemic clamp.

SECONDARY OUTCOMES:
Changes in macrovascular function | One week
  Macrovascular function will be assessed with flow-mediated dilation
Changes in microvascular function | One week
  Macrovascular function will be assessed with EndoPAT
Changes in cognitive abilities | One week
  Cognitive computer tests performed during study
Changes in circadian rhythms | One week
  Salivary dim-light melatonin offset will be assessed
Changes in metabolic tissue function | One week
  Tissue biopsies will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Josiane L. Broussard, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Full list of publications — http://www.ncbi.nlm.nih.gov/sites/myncbi/1JaM6qKzqsa5p/bibliography/45302103/public/?sort=date&direction=ascending